CLINICAL TRIAL: NCT02616172
Title: Safety of Infusion of Autologous Human Bone Marrow Mononuclear Fraction in Children With Sensorineural Hearing Loss
Brief Title: Autologous Bone Marrow Harvest and Transplant for Sensorineural Hearing Loss
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Restructuring Cell Lab
Sponsor: James Baumgartner, MD (Other)
Responsible Party: Sponsor-Investigator, James Baumgartner, MD, Primary Investigator, AdventHealth
Organization: AdventHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 695389
Record Dates: First submitted 2015-08-19; First posted 2015-11-26 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous bone marrow infusion (Experimental): One time administration of autologous bone marrow mononuclear cells intravenously, minimum dose of 6 million cells per kg Total nucleated cells.
  Interventions: Genetic: Autologous Bone Marrow Infusion

INTERVENTIONS:
Genetic: Autologous Bone Marrow Infusion — The subjects autologous bone marrow cells harvested at Florida Hospital will be infused intravenously by gravity
  Other Names: Cell based therapy

SUMMARY:
Autologous human bone marrow mononuclear fraction (BMMF) will be harvested and given to children with bilateral moderate to severe sensorineural hearing loss. The aim is to determine if bone marrow mononuclear fraction (BMMF) infusion is safe, feasible, improves inner ear function, audition, and language development.

DETAILED DESCRIPTION:
Autologous human bone marrow mononuclear fraction (BMMF) will be given to children with bilateral moderate to severe sensorineural hearing loss.

Subjects will come to Orlando for pretesting to include an Magnetic Resonance Imaging (MRI), Auditory brainstem response (ABR), blood work: Complete metabolic panel (CMP), Complete blood count (CBC), Hepatic Function Panel, Prothrombin (PT), Partial thromboplastin time (PTT), International normalized ration (INR), Chest Xray, and a Speech and Language Evaluation.

After pretesting, the subjects will undergo a bone marrow harvest and then receive their autologous bone marrow mononuclear fraction (BMMF) intravenously. The subjects will then be monitored for 24 hours post infusion. After 24 hours, the subject will undergo repeat blood work and a chest x ray. Subjects will then be discharged home. Subjects will follow up in Orlando at 1 month, 6 months and 1 year post infusion. Follow up testing will repeat the exams performed at pretesting.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of sensorineural hearing loss that is,

   * Bilaterally Moderate or Profound in degree
   * Symmetrical or asymmetrical configuration
   * Sudden or progressive in presentation
2. Normally shaped cochlea, as determined by Magnetic Resonance Imaging or computed tomography (CT)
3. The loss must be considered:

   * Acquired
   * Unknown with genetic testing negative. (Genetic testing is not required for Cytomegalovirus (CMV) positive children due to Cytomegalovirus (CMV) known to be number one cause of hearing loss)
4. Fitted for hearing aids no later than six months post detection of loss unless not recommended by treating audiologist or physicians
5. Enrollment in a parent/child intervention program
6. Age 2 years - 6 years old at time of infusion with 2 to 4 years of time elapsed since diagnosis of hearing loss at the time of bone marrow mononuclear fraction (BMMF) infusion.
7. Ability of the child and caregiver to travel to Orlando, and stay for at least 4 days, and to return for all follow-up visits.

Exclusion Criteria:

1. Inability to obtain all pertinent medical records:

   * (pertinent physician notes, speech language pathology notes, laboratory findings, test results and imaging studies-must be sent to the research team at least prior to the subject arriving at the study location for preliminary screening and eligibility assessment, preferably14 days before the scheduled visit.)
2. Known history of:

   * Recently treated (ear or any infections) infection less than 2 weeks before infusion.
   * Renal disease of altered renal function as defined by serum creatinine > 1.5 mg/dl at admission.
   * Hepatic disease or altered liver function as defined by Alanine Transaminase (SGPT) > 150 U/L, and or Total Bilirubin > 1.3 mg/dL
   * Malignancy
   * Immunosuppression as defined by White Blood Cell (WBC) < 3,000 at admission
   * Human Immunodeficiency Virus (HIV)
   * Hepatitis B
   * Hepatitis C
   * Pneumonia, or chronic lung disease requiring oxygen
3. Any evidence of active maternal infection during the pregnancy
4. Participation in a concurrent intervention study
5. Mild hearing loss with no evidence of moderate of severe loss
6. Unwillingness or inability to stay for 4 days following infusion (should problems arise following the infusion) and to return for the one month, six month and one year follow-up visits.
7. Evidence of conductive hearing loss
8. Documented recurrent middle ear infections which are frequent (>5 per year)
9. Otitis media at the time of examination
10. Before 2 years from identification of hearing loss at time of infusion
11. After 4 years from identification of hearing loss at time of infusion
12. Diagnosis of the following syndromic cause for hearing loss

    * CHARGE
    * Waardenburg
    * Brachio-Oto-Renal
    * Pendred
    * Alport
    * Treacher-Collins
    * Usher
    * Stickler Syndrome

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
physiological parameter: Blood Pressure | Change from baseline to 24 hours after stem cell infusion
  Assessing change from baseline systolic blood pressure to post stem cell infusion systolic blood pressure. The metric for summarizing measurements is millimeters of mercury.
physiological parameter: Pulmonary Endothelial Damage | Change from baseline to 24 hours post infusion
  Measured by the number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Change: Number of Participants With Treatment-Related Adverse Events as Assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 for Hepatic Injury | Change from baseline to post infusion day 1
  The reticuloendothelial system can sequester immature blood elements, theoretically resulting in hepatic injury. An acute elevation of the aspartate transaminase (AST) and Alanine Aminotransferase test (ALT) hepatic enzymes >5.0 - 20.0 x upper limit normal (ULN) in the first 24 hours post infusion will trigger the stopping rules. This level corresponds to the Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0 Grade 3 adverse event. It is unlikely that "end vessel" microthrombosis would occur in the liver due to the dual blood supply of the liver and the lung is the first pass organ. This will be reported as the number of participants with abnormal laboratory values and adverse events related to treatment.
Change: Number of Participants With Treatment-Related Adverse Events as Assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 for Neurological status | Change in baseline to 1 day post infusion
  Change in the subject's acute neurologic status will be monitored hourly for 4 hours after infusion. Data recorded include Glasgow Coma Scale (GCS) from infusion to discharge. Grade 3 Central Nervous System (CNS) event as defined in the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0 occurring within 12 hours of cellular product infusion will trigger the stopping rules. Other changes temporally related to infusion (those events occurring within 12 hours of infusion) will be considered associated with the protocol and recorded as an adverse event. This will be reported as the number of participants with adverse events related to treatment.
Incidence of Treatment-Emergent Adverse Events for Pulmonary Status | Baseline to 24 hours after infusion
  Blood-oxygen saturation will be monitored by finger oximeter. Moderate respiratory dysfunction within the first 24 hours post infusion will be considered an adverse event but will not warrant stopping the trial unless recommended by the Data Safety Monitoring Board. In the event of pulmonary dysfunction, standard supportive therapy will be given. Pulmonary symptoms/events corresponding to the Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 Grade 3 will trigger the stopping rules

SECONDARY OUTCOMES:
Auditory Brainstem Response | Baseline, 1 month, 6 months, and 1 year
  Audiometry, to-acoustic emissions and Auditory Brainstem Response will be used to assess the physiologic integrity of the neural structures which are critical to normal audition and speech. Changes in these areas will be evaluated by repeating the measures all follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: James Baumgartner, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital for Children, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided